CLINICAL TRIAL: NCT01426555
Title: FES-Rowing Versus Zoledronic Acid to Improve Bone Health in SCI: A Comparative Clinical Trial
Brief Title: FES-Rowing Versus Zoledronic Acid to Improve Bone Health in Spinal Cord Injury (SCI)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Incomplete data set & analysis
Sponsor: Antonio Lazzari (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Spaulding Rehabilitation Hospital (Other); VA Boston Healthcare System (U.S. Federal Agency); Massachusetts General Hospital (Other)
Responsible Party: Sponsor-Investigator, Antonio Lazzari, PI, Boston VA Research Institute, Inc.
Organization: Boston VA Research Institute, Inc. (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 109241
Record Dates: First submitted 2011-06-08; First posted 2011-08-31 (Estimated); Results first posted 2016-03-10 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-03

CONDITIONS: Osteoporosis
Keywords: Disorder of Bone Density and Structure, Unspecified; Weakening of the bone structure
MeSH Terms: conditions — Osteoporosis | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FES Rowing (Active Comparator): Group 1 - FES-Rowing Exercise for entire study period
  Interventions: Other: FES-Rowing
- FES Rowing + Zoledronic acid (Experimental): Group 2 - FES-Rowing Exercise for entire study period plus Zoledronic Acid 5mg administered by i.v. infusion one-time at the end of observation period
  Interventions: Other: FES-Rowing; Drug: Zoledronic acid

INTERVENTIONS:
Other: FES-Rowing — FES- Rowing Exercise
  Other Names: Rowing exercise
Drug: Zoledronic acid — 5 mg IV single dose
  Other Names: Reclast
  Arms: FES Rowing + Zoledronic acid

SUMMARY:
This is a research study to determine the effects of functional electrical stimulation (FES) rowing and a drug called zoledronic acid in bone health. The investigators hoped to learn if zoledronic acid treatment will increase bone mineral density in persons with chronic spinal cord injury (SCI) who received it. The investigators also want to find out if zoledronic acid is safe for persons with SCI to take without causing too many side effects.

DETAILED DESCRIPTION:
This research study was designed to determine the effects of functional electrical stimulation (FES) rowing and a drug called zoledronic acid in bone health in individuals who have suffered a spinal cord injury (SCI). The investigators hoped to learn if zoledronic acid treatment would increase bone mineral density in persons with chronic spinal cord injury. This was designed and conducted as a three center study with multiple investigators. The investigators also had a goal to find out if zoledronic acid is safe for persons with SCI without causing too many side effects.

The Prime recipient of funding is Spaulding Rehabilitation Hospital (SRH). Dr. Leslie Morse is the Principal Investigator for the study, the coordination of the study was located at Spaulding Rehabilitation Hospital. Through a sub-award a research group from the Veterans Administration of Boston Healthcare System was contracted to conduct DXA scans, blood draws and zoledronic acid administration to support this study. Through another sub-award from SRH, another Investigator from Massachusetts General Hospital (MGH) participated conducting CT scans for the study. All adverse events related to this study were to be monitored and recorded by investigators at SRH.

Seventy subjects age 18 years or older and wheelchair dependent at least 50% of the time because of an SCI were enrolled. Enrollment and initial screening for the study and follow up was performed at SRH. After enrollment the subjects were randomized to 1) FES-rowing alone or 2) FES-rowing plus a 1-time infusion of zoledronic acid. Following a variable period of strength training which was necessary for preparing quads and hamstrings for extended FES use, enrolled participants were planned to begin a regular rowing program for 12 months at the Cardiovascular Laboratory at the Spaulding Rehabilitation Hospital . DXA scans to measure bone mineral density were planned to be performed at the VA Boston Healthcare System-Jamaica Plain Campus (VABHS) three times during the study on all participants. In addition, 25 subjects in each arm of the study were planned to receive CT scans of their knees at MGH at the beginning and end of the study. Up to 20 subjects were to have an additional CT scan (at MGH) six months into rowing. Research blood samples were planned to be collected at VABHS five times during duration of the study and stored at the VA for further study of molecular markers of bone turnover. All participants were expected to be screened for renal function and calcium and vitamin D levels at the beginning and end of the study, with additional renal screening done before and after the zoledronic acid infusion. Calcium and vitamin D supplements were to be provided to each subject throughout the study. Those with insufficient vitamin D levels were to be provided additional repletion and planned to be periodically rechecked. Up to 15 male subjects were asked to have two echocardiograms at one of the SRH sites - one at the beginning of the study and the other halfway through the year-long rowing regimen.

ELIGIBILITY:
Inclusion Criteria:

* male and female SCI outpatients
* women of child bearing age will be required to use an acceptable birth control method throughout the study
* aged 18 - over the age of 40
* physician's cardiac clearance to exercise
* who were at least age 14 at time of injury
* who are at least 18 months post injury
* who have a C4 spinal cord injury or lower

Exclusion Criteria:

* initial blood pressure higher than 140/90
* patients with orthostatic hypotension
* an active grade 2 or greater pressure ulcers
* lower extremity contractures
* history of significant arrhythmias
* coronary disease
* diabetes
* neurological or renal disease
* cancer
* other neurological disease (i.e. stroke, peripheral neuropathy, myopathy)
* any implanted electronic device
* active treatment for epilepsy
* recent weight change
* regular use of tobacco
* family history of arrhythmia or sudden cardiac death
* current use of cardioactive or antidepressant medications
* current use of medications that may affect fracture risk including:
* bisphosphonates
* PTH and PTH analogs
* androgenic steroids
* estrogenic steroids
* glucocorticoids
* antiepileptics
* lithium.
* Any subject with a planned invasive dental procedure will be excluded.

These criteria will be reviewed by telephone survey followed by a health exam where blood pressure will be assessed and a skin and neurological exam performed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Morse, DO, Principal Investigator — Spaulding Rehab. Hospital; Antonio A Lazzari, MD, Principal Investigator — Boston Division VAMC - New England
Locations (2):
- United States (2):
  - Boston VAMC, Boston, Massachusetts
  - Spaulding Rehab. Hospital, Charlestown, Massachusetts

IPD SHARING:
Plan to Share IPD: No
The study has been closed by the VABHS IRB.

RESULTS

PARTICIPANT FLOW:
Groups:
- Rowing Arm: Prior to FES-row, subjects undertook a 2 -12 weeks strength-training program at SRH, depending on how the subjects respond to the FES-strength training. Subjects who completed strength training, progressed to rowing.
  In the FES-Rowing program, the goal was for each subject to achieve an exercise intensity of 75-85% maintained for a continuous 40 minutes performed 3 times each week in additional to maintaining strength training at home on days when they are not rowing.
  All subjects received a daily minimum supplementation of 1000mg Calcium & 1000 IUs of Vitamin-D supplementation during the duration of the program.
- ZA Infusion Arm: Prior to FES-row, subjects undertook a 2 -12 weeks strength-training program at SRH, depending on how the subjects respond to the FES-strength training. Subjects who completed strength training, progressed to rowing.
  In the FES-Rowing program, the goal was for each subject to achieve an exercise intensity of 75-85% maintained for a continuous 40 minutes performed 3 times each week in additional to maintaining strength training at home on days when they are not rowing.
  After the observation period, subjects in the FES rowing plus zoledronic acid arm were planned to receive Zoledronic Acid (Reclast ®) administered as a dose of 5mg intravenously.
  All subjects received a daily minimum supplementation of 1000mg Calcium & 1000 IUs of Vitamin-D supplementation during the duration of the program.
Period: Overall Study
Arm/Group | Rowing Arm | ZA Infusion Arm
Started | 35 | 35
Completed | 17 | 20
Not Completed | 18 | 15

BASELINE CHARACTERISTICS:
Groups:
- ZA Infusion Arm: Thirty five subjects in each arm, age 18 years or older and wheelchair dependent at least 50% of the time because of an SCI were enrolled.
- Rowing Arm: Thirty five subjects, in each arm age 18 years or older and wheelchair dependent at least 50% of the time because of an SCI were enrolled.
- Total: Total of all reporting groups
Arm/Group | ZA Infusion Arm | Rowing Arm | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 35 | 70
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 37.2 [20.7 to 63.5] | 39.0 [21.1 to 65.0] | 38.1 [20.7 to 65.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 32 | 32 | 64
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Improvement of Bone Mass as Measured by Sequential Evaluation of Bone Density and Bone Structure
Description: This work was designed to determine if FES-rowing plus Zoledronic acid is superior to FES-rowing alone reversing deterioration and weakening of the bones due to SCI and was planned to confirm the effects of FES-rowing in bone structure in patients not receiving Zoledronic Acid.
Time Frame: 12 months
Population: Data was never analyzed because the study was closed by the VABHS IRB. Full dataset is unavailable for analysis.
Groups:
- ZA Infusion Arm: Thirty Five subjects in each arm, age 18 years or older and wheelchair dependent at least 50% of the time because of an SCI were planned to be enrolled.
  No Data was analyzed because dataset is not available to VABHS Study team.
- Rowing Arm: Thirty Five subjects, in each arm age 18 years or older and wheelchair dependent at least 50% of the time because of an SCI were planned to be enrolled.
  No Data was analyzed because dataset is not available to VABHS Study team.
Arm/Group | ZA Infusion Arm | Rowing Arm
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Validation of DXA Scanning in Patients With SCI
Description: This study has been designed to evaluate whether sequential DXA scanning of the distal femur and proximal femur is an appropriate clinical tool to monitor bone changes in response to either treatment. Evaluation of bone density by DXA was planned to be compared to CT scans of the distal femur and proximal tibia.
Time Frame: 12 months
Population: Dataset unavailable for analysis to VABHS study team. The study was closed by the VABHS IRB.
Groups:
- ZA Infusion Arm: Thirty Five subjects in each arm, age 18 years or older and wheelchair dependent at least 50% of the time because of an SCI, were enrolled.
  Dataset unavailable for analysis to VABHS study team. The study was closed by the VABHS IRB.
- Rowing Arm: Thirty Five subjects, in each arm age 18 years or older and wheelchair dependent at least 50% of the time because of an SCI, enrolled.
  Dataset unavailable for analysis to VABHS study team. The study was closed by the VABHS IRB.
Arm/Group | ZA Infusion Arm | Rowing Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were followed up for the duration of the study for up to 4 years.
Description: Adverse Events data not complete on participants to the IND Sponsor.
Groups:
- ZA Infusion Arm: No adverse event data were available for the remaining 9 participants.
- Rowing Arm: No adverse event data were available for the remaining 16 participants.
Arm/Group | ZA Infusion Arm | Rowing Arm
Serious Adverse Events (participants affected / at risk) | 6/26 | 6/19
Other Adverse Events (participants affected / at risk) | 15/26 | 15/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZA Infusion Arm (N=26) | Rowing Arm (N=19)
UTI (Renal and urinary disorders) | 2 (2) | 1 (1) — Hospitalized for UTI unrelated to rowing.
Kidney Stone (Renal and urinary disorders) | 1 (1) | 1 (1) — Kidney stone
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Fractured bone. Patient withdrew from the study before underdoing study procedures.
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) — Subject developed a Upper Respiratory Tract Infection
Elevated Heart Rate (Cardiac disorders) | 0 (0) | 1 (2)
High Fever (Infections and infestations) | 1 (1) | 1 (1) — High Fever, vomiting, chills and fatigue.
Pressure Ulcers (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZA Infusion Arm (N=26) | Rowing Arm (N=19)
Spasticity (Musculoskeletal and connective tissue disorders) | 5 (10) | 2 (2) — Spasms or contractions.
Fatigue / Not Feeling Well / Asthenia (General disorders) | 6 (13) | 6 (20) — Fatigue, Not Feeling Well, Asthenia, Dizziness
Injury / Skin Cuts (Injury, poisoning and procedural complications) | 3 (11) | 2 (2) — Injury, skin cuts, bruises
Fracture (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) — Fracture
Blood Pressure (Cardiac disorders) | 4 (6) | 2 (8) — High Blood Pressure Low Blood Pressure
Gastrointestinal Disorders (Gastrointestinal disorders) | 5 (5) | 7 (14) — gastroenteritis, stomach pain, constipation or diarrhea.
Cardiac Conditions / Arrhythmias (Cardiac disorders) | 3 (7) | 4 (5) — Fast heart rate, atrial fibrillation, arrhythmias
Respiratory Illness/Disorder (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 5 (9) — Respiratory Illness/Disorder, Bronchitis, Upper respiratory infection, Flu symptoms
Pain / Aches / Neuralgia (Musculoskeletal and connective tissue disorders) | 8 (29) | 9 (24) — Aches Pain Neuralgia including musculoskeletal pains
Fever (General disorders) | 5 (5) | 3 (3) — fever, chills
Falls / Injuries (Injury, poisoning and procedural complications) | 10 (11) | 8 (11) — fall or injury car accident with injury
Pressure Ulcer / Sore (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4) — Pressure Ulcer / Sore Decubitus Ulcer
Urinary Tract Infection (Renal and urinary disorders) | 5 (7) | 6 (11) — urinary tract infections
Autonomic Dysreflexia / Other General Symptoms (General disorders) | 5 (12) | 8 (10) — autonomic dysreflexia, other general symptoms

LIMITATIONS AND CAVEATS:
No Data Safety Monitor Board established for this project. Incomplete data set and analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No